CLINICAL TRIAL: NCT03843008
Title: Role of Melatonin in the Acute Phase of Stroke as Measured by Interleukin 6 Biomarker
Brief Title: Melatonin in Acute Stroke
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study never started
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB201801934
Record Dates: First submitted 2019-02-13; First posted 2019-02-15 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Stroke, Acute; Ischemic Stroke
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — Melatonin

STUDY DESIGN:
Intervention Model Description: Patients will receive 3mg of melatonin or no melatonin for up to seven days or for the duration of his or hospital stay for a maximum total of 21mg of melatonin.
Who Masked: Participant, Investigator
Masking Description: At discharge, the patient will be assessed via a blinded-physician for NIHSS and this value will be recorded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melatonin Group (Experimental): Participants will receive 3mg of melatonin at 18:00 (+/- one hour) each evening up to seven days or for the duration of his or her hospital stay.
  Interventions: Dietary Supplement: Melatonin
- No Melatonin Group (No Intervention): Participants will receive no melatonin for the length of their hospital stay.

INTERVENTIONS:
Dietary Supplement: Melatonin — Participants in the Melatonin Group will receive 3mg of melatonin each evening for up to seven days for a maximum total of 21mg of melatonin.
  Other Names: Nature Made melatonin; N-acetyl-5-methoxytryptamine
  Arms: Melatonin Group

SUMMARY:
This study will measure Interleukin 6 (IL-6), a well-documented inflammatory biomarker that is increased in the acute phase of stroke, and to compare its levels after the administration of melatonin - a well-documented anti-inflammatory and anti-oxidant - that regulates circadian rhythm, which helps promote sleep.

DETAILED DESCRIPTION:
Stroke is a major cause of debilitation in the first world, with few therapeutic options when it comes to improvement in quality of life and morbidity, besides physical and occupational therapy. It affects people of all nationalities, creeds, and socioeconomic classes through a narrow array of mechanisms. With all those mechanisms, a common outcome is shared: derangement of the brain parenchymal architecture. This derangement is non-selective in its destruction with obscuration of the blood brain barrier and the glymphatic system, and with bleeding as a common sequela; the oxidative stress of the hemoglobin-heme-iron compound causing further injury. This study will measure Interleukin 6 (IL-6), a well-documented inflammatory biomarker that is increased in the acute phase of stroke, and to compare its levels after the administration of melatonin - a well-documented anti-inflammatory and anti-oxidant - that regulates circadian rhythm, which helps promote sleep. Any increased time spent in a restful state because of melatonin increases the clearance of waste products after a catastrophic event, like in stroke.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted to the Neuroscience Critical Care Unit with a confirmed ischemic stroke
* Patients with a clinical history and examination consistent with an ischemic stroke (stroke must be confirmed by a brain CT and/or MRI scan)
* Eligible patients will have been treated with TPA and/or thrombectomy.

Exclusion Criteria:

* Prisoners
* Patients with severe cognitive impairment and/or aphasia (if no family member is available to sign consent)
* Recent (<1 month) infection
* Pregnant females

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Change in serum Interleukin 6 (IL 6) | Baseline, Week 1
  Determine whether Interleukin 6 (IL-6) is lowered after the administration of melatonin. At 6:00 (+/- one hour) each morning for the duration of the hospital stay, patient will have IL-6 biomarker assayed. This testing will continue for the duration of the hospital stay, or for seven days (whichever comes first).

CONTACTS AND LOCATIONS:
Overall Officials: Andreja Packard, MD, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida College of Medicine-Jacksonville, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No